CLINICAL TRIAL: NCT03100214
Title: Effects of an Early Rehabilitation Program During Hospitalization in Adolescents and Adults Patients With Cystic Fibrosis: Randomized Clinical Trial
Brief Title: Effects of an Early Rehabilitation Program During Hospitalization in Patients With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 150443
Record Dates: First submitted 2017-01-31; First posted 2017-04-04 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Patients randomized to the control group will continue to receive the physiotherapeutic follow-up performed by the physiotherapist of the Program for Adults with CF during the hospitalization period. Supervision includes respiratory physiotherapy involving inhalation therapy and techniques for removal of secretions.
  Interventions: Other: Control
- Exercise (Experimental): Patients randomized to the intervention group, in addition to routine physical therapy follow-up, will receive an early rehabilitation program, which will begin within the first 48 hours after admission. The patient will perform physical training (aerobic and anaerobic) 5 times a week during the hospitalization period, with sessions about an hour. The professional who supervises the training will be blinded to the results of the measurements.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Patients randomized to the intervention group, in addition to routine physical therapy follow-up, will receive an early rehabilitation program, which will begin within the first 48 hours after admission. The patient will perform physical training (aerobic and anaerobic) 5 times a week during the hospitalization period, with sessions about an hour. The professional who supervises the training will be blinded to the results of the measurements.
  Arms: Exercise
Other: Control — Patients randomized to the control group will continue to receive the physiotherapeutic follow-up performed by the physiotherapist of the Program for Adults with CF during the hospitalization period. Supervision includes respiratory physiotherapy involving inhalation therapy and techniques for removal of secretions
  Arms: Control

SUMMARY:
Studies demonstrate that exercise increases the maximal oxygen uptake, peak oxygen consumption, reduce effort-induced lactic acid production, and increase skeletal muscle oxidative capacity, as well as psychological aspects such as increased self-esteem and improvement of the quality of life.

In the literature there is only one study involving rehabilitation in hospitalized pediatric patients with cystic fibrosis. Thus, more information on in-hospital rehabilitation is required in adult cystic fibrosis patients.

The present study aims to evaluate the effects of an early rehabilitation program, based on aerobic training and muscle strength training, in adolescent and adult patients with cystic fibrosis hospitalized at Hospital de Clinicas de Porto Alegre for exacerbation of lung disease.

DETAILED DESCRIPTION:
After completing the study inclusion criteria, the individual will be invited to participate and will receive the consent form for signature.

The patient will be submitted to the following evaluations: quality of life questionnaire for cystic fibrosis, spirometry, Shwachman-Kulczycki score, modified dyspnea questionnaire (Modified Medical Research Council), maximum repetition test, six minute walk test and blood sample for the determination of inflammatory markers. These evaluations should be performed within the first 48 hours of hospitalization, and will be repeated on the last day of hospitalization.

In the period up to 48 hours after hospital admission, patients will be randomized to either the intervention group or the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 16 years and older,
* Regularly followed up in the Hospital de Clinicas de Porto Alegre Program for Adolescents and Adults with Cystic Fibrosis with a diagnosis of cystic fibrosis confirmed according to the consensus criteria,
* Admitted to hospital admission due to exacerbation of lung disease.
* Hospital stay will be defined as the stay equal to or greater than 24 hours in any Hospital de Clinicas de Porto Alegre unit.

Exclusion Criteria:

* Patients with cardiac, orthopedic or trauma complications that make it impossible to perform the proposed exercises;
* Pregnant patients;
* Patients with hemodynamic instability, massive hemoptysis, pneumothorax, and continuous use of noninvasive ventilation.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2016-08; Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Distance walked during the six minute walk test | up to 14 days
  The six-minute walk test will be performed at hospital discharge.

SECONDARY OUTCOMES:
Forced expiratory volume in the first second | up to 14 days
  The spirometry will be performed at hospital discharge.
Cystic fibrosis quality of life questionary | up to 14 days
  Cystic fibrosis quality of life questionary will be performed at hospital discharge.
C-reative protein | up to 14 days
  C-reative protein will be performed at hospital discharge.
Interleukin-6 | up to 14 days
  Interleukin-6 will be performed at hospital discharge.
Interleukin-8 | up to 14 days
  Interleukin-8 will be performed at hospital discharge.
Tumor necrosis factor | up to 14 days
  Tumor necrosis factor will be performed at hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo de Tarso R Dalcin, PhD, Study Director — Hospital de Clínicas de Porto Alegre
Locations (1):
- Paulo de Tarso Dalcin, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided